CLINICAL TRIAL: NCT04874792
Title: Clinical Characteristics of Deceased With COVID-19: Review of Medical Records in a Referral Hospital Dedicated for COVID-19
Brief Title: Clinical Characteristics of Deceased With COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Mohammad Mahfuzul Hoque, Assistant Professor, Dhaka Medical College
Other Study IDs: ERC-DMC-ECC/2020/142
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: COVID19; Clinical Characteristics; Deceased
MeSH Terms: conditions — COVID-19; Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe the clinical characteristics of patients who died from COVID-19 in the largest hospital in Bangladesh to understand the risk associated with COVID-19 related mortality in this region. This is a retrospective study where a review of hospital records of patients will be done who died from COVID-19 in Dhaka Medical College Hospital from 3rd May to 31 August 2020. All available demographic, clinical, laboratory information, radiological feature, and patients' management will be retrieved from the record section to be analyzed and described.

DETAILED DESCRIPTION:
In this retrospective observational study, every consecutive patient who died and tested positive for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in Dhaka Medical College Hospital from 2nd May 2020 to 31 August 2020 were included. The paper files of patients were retrieved from the record section of the hospital as only a paper-based recording is maintained in the hospital. Patients with suspected COVID-19 were excluded from the study who tested negative for Reverse Transcriptase Polymerase Chain Reaction (RT PCR for SARS-CoV-2).

A preformed case record form (CRF) was used to collect all available demographic, clinical information including presentation, investigation, and treatment from hospital paper file from the record section. The severity of disease for COVID-19 was classified according to National Guidelines on Clinical Management of COVID-19 Version 8.0, 5 November 2020. The mild disease was defined as an individual with COVID-19 with prodromal symptoms without dyspnea and radiological abnormality. The moderate disease was defined as abnormal chest imaging with the saturation of oxygen ≥ 90% and severe disease was denied as saturation of oxygen less than 90%. All data were summarized, analyzed with SPPS 26.

RT PCR for SARS-CoV-2 assay is done in the virology department of Dhaka Medical College to detect SARS-Cov-2 RNA from samples taken from suspected patients. Nasopharyngeal swabs and the oropharyngeal swab were taken from patients. Biochemical, hematological investigations are done in the clinical pathology department of the hospital and paper reports are sent to respective patients' files. Laboratory measurements were collected for analysis which is available in the file of deceased patients in the record section.

ELIGIBILITY:
Inclusion Criteria:

* All Patients died from COVID-19 confirmed with rt PCR for SARS-CoV-2

Exclusion Criteria:

* Suspected COVID-19 patients negative for rt PCR for SARS-CoV-2 and
* Age less than 14 year

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients died from COVID-19 in Dhaka Medical College Hospital confirmed by Real-Time reverse transcription Polymerase Chain Reaction during the period from 3rd May 2020 to 31st August 2020.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Characteristics | 03/05/2020 to 31/08/20
  Demography, Clinical presentation, Treatment

SECONDARY OUTCOMES:
Duration from admission to death | 03/05/2020 to 31/08/20
  Duration of Hospitalization from admission to death in different comorbidity and disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad M Hoque, FCPS, Principal Investigator — Assistant Professor of Medicine, Dhaka Medical College
Locations (1):
- Dhaka Medical College Hospital, Dhaka, Bangladesh